CLINICAL TRIAL: NCT05298839
Title: Effect of COVID-19 Infection on the Performance of Adolescent Professional Overhead Athletes
Acronym: Atılım Unv
Status: Completed | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Other Study IDs: E-59394181-604.01.02-13774
Record Dates: First submitted 2022-03-25; First posted 2022-03-28 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Sport Performance, Professional Overhead Athletes
Keywords: COVID-19; sport performance; adolescent athletes; overhead sport
MeSH Terms: conditions — COVID-19 | interventions — Hand Strength; Reaction Time; Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19
  Interventions: Diagnostic Test: Evaluation of core muscle endurance, hand grip strength, upper extremity functional performance, reaction time, agility performance and 3 minutes step test
- Non COVID-19
  Interventions: Diagnostic Test: Evaluation of core muscle endurance, hand grip strength, upper extremity functional performance, reaction time, agility performance and 3 minutes step test

INTERVENTIONS:
Diagnostic Test: Evaluation of core muscle endurance, hand grip strength, upper extremity functional performance, reaction time, agility performance and 3 minutes step test — Core muscle endurance was evaluated with extensor muscle endurance test, flexor muscle endurance test and lateral muscle endurance test.
  Hand Grip Strength was evaluated with Jamar hand dynamometer. Upper extremity functional performance was evaluated with health ball throwing test.
  Reaction time was evaluated with Fitlight Trainer. Agility performance was evaluated with Pro-agility test. Cardiovascular endurance was evaluated with the 3-minute step test.

SUMMARY:
COVID-19 is known to also cause damage outside the pulmonary system, particularly the cardiovascular and the musculoskeletal system. The studies on the effects of COVID-19 infection on different populations may provide valuable information for health professionals. Derangements in the cardiorespiratory and musculoskeletal systems which normally direct effect on the sports performance of athlete together with physical inactivity during COVID-19 infection are the main factors that may decrease the performance of the professional athletes. Although it may be well anticipated that COVID-19 will reduce sports performance; there are scarce studies in the literature. The aim of this study is to compare the sports performance of adolescent athletes that has COVID-19 infection with those did not.

DETAILED DESCRIPTION:
Extensor muscle endurance, flexor muscle endurance and the lateral core muscle endurance were evaluated. All tests were performed by a chronometer and test was terminated as the position was lost and the time passed was recorded. Hand grip strength was measured by Jamar hand dynamometer. Health ball throwing test was used to evaluate upper extremity open kinetic chain and explosive power. Pro-agility test was used to evaluate the agility. Step test was performed for 3 minutes with a 30 cm high step board.

ELIGIBILITY:
Inclusion Criteria:

* Basketball, volleyball, handball, tennis and American football players
* Between 12 to 20
* Performing sports-specific training more than two times a week at least for 1 year

Exclusion Criteria:

* Vertebral, upper or lower extremity injury within the last 6 weeks or had undergone a surgery

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Professional athletes
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Core Muscle Endurance | June 2021- August 2021
  Four different tests were used to evaluate core stabilization. Sorensen test was performed for extensor muscle endurance. For the Sorensen test, young athletes were laid supine in a fixed bed of 76 cm height and 61 cm width; and asked to extend their body over the pelvis and keep the position as long as they could. Core flexor muscle endurance was measured in the position of body flexion of 60°, and knee and hip flexion of 90° and athletes were asked to keep the position as long as possible. To evaluate the general core muscle power, young athletes were asked to lie prone and lift their body on forearm and toes and keep the position as long as possible. For the lateral core muscle endurance athletes were asked to get into left and right decubitus position respectively and lift their body on forearm and toes and keep the position as long as possible. All tests were performed by a chronometer and test was terminated as the position was lost and the time passed was recorded
Jamar hand dynamometer | June 2021- August 2021
  Hand grip strength was measured by Jamar hand dynamometer. Measurement was taken three times for both right and left sides while the subject was sitting on a chair, shoulder in adduction and elbow at 90 degree flexion. Twenty seconds of rest was given between the two measurements. Mean value of three results were calculated and recorded as kPa
Upper Extremity Functional Performance | June 2021- August 2021
  Health ball throwing test was used to evaluate upper extremity open kinetic chain and explosive power. Subjects were told to hold the 3 kg health ball and throw it horizontally to the furthest possible point using two hands. The distance between the starting point and the first contact point on the floor was recorded as centimeters. Test was repeated three times and mean values were recorded.
Reaction Time | June 2021- August 2021
  Reaction time and dynamic postural control was evaluated with ''Fitlight TrainerTM'' (Fitlight Trainer Corporation, Thensvej, Risskov, Denmark). Athletes were asked to turn out the LED lights placed on the wall that were randomly turned on and the total number of the LED lights they turned off and their reaction time were noted as seconds
Agility Performance | June 2021- August 2021
  Agility test was used to evaluate the agility. Markers were placed at the left and right side 5 yard (4,57 m.) away from the starting point. Photocell gate was placed at the starting point to detect the passing times of the athletes. Athletes took position at the starting point and they were told to touch the right marker and then the left marker and turn back to starting point
3 Minutes Step Test | June 2021- August 2021
  A step board with the height of 30 cm., oxygen saturation probe, pulse oximeter, metronome and chronometer were used for the test. Athletes were informed about the test and rhythm of the metronome was delivered for certain time to get used to the rhythm. Athletes started the test with the foot they preferred and were asked to step on and off the board in harmony with the rhythm of the metronome. Oxygen saturation, pulse rates and Modified Borg Scale score that is used to identify fatigue were recorded at the end of the test

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)